CLINICAL TRIAL: NCT03555071
Title: A Double-blind, Randomized, Bridging Clinical Trial to Evaluate the Consistency, Immunogenicity and Safety of Live Attenuated Varicella Vaccines for Children
Brief Title: A Phase 3 Lot-consistency Clinical Trial of Live Attenuated Varicella Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-VZV-3002
Record Dates: First submitted 2018-04-16; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-04

CONDITIONS: Varicella
Keywords: live attenuated varicella vaccine; consistency; immunogenicity; safety; children
MeSH Terms: conditions — Chickenpox

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group1 (Experimental): The investigated vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd at commercialized scale.
  Intervention: Live attenuated varicella vaccine manufactured at commercialized scale
  Interventions: Biological: Vaccine manufactured at commercialized scale
- Experimental Group2 (Experimental): The investigated vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd at commercialized scale.
  Intervention: Live attenuated varicella vaccine manufactured at commercialized scale
  Interventions: Biological: Vaccine manufactured at commercialized scale
- Experimental Group3 (Experimental): The investigated vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd at commercialized scale.
  Intervention: Live attenuated varicella vaccine manufactured at commercialized scale
  Interventions: Biological: Vaccine manufactured at commercialized scale
- Control Group (Active Comparator): The control vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd at trial-scale.
  Intervention: Live attenuated varicella vaccine manufactured at trial-scale
  Interventions: Biological: Vaccine manufactured at trial-scale

INTERVENTIONS:
Biological: Vaccine manufactured at commercialized scale — Single subcutaneous injection of the investigated live attenuated varicella vaccine (0.5 ml) on Day 0
  Arms: Experimental Group1; Experimental Group2; Experimental Group3
Biological: Vaccine manufactured at trial-scale — Single subcutaneous injection of the control live attenuated varicella vaccine (0.5 ml) on Day 0
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate consistency, immunogenicity and safety of live attenuated varicella vaccines manufactured at commercialized scale in aged 1-3 years children.

DETAILED DESCRIPTION:
The study is a single-center, double-blind, randomized, bridging clinical trial. The purpose of this study is to evaluate the consistency between each two lots of live attenuated varicella vaccines, to evaluate the non-inferiority of the immunogenicity of live attenuated varicella vaccines manufactured at commercialized scale compared to trial-scale, and to evaluate the safety of live attenuated varicella vaccines. 1197 healthy Chinese children aged 1 to 3 years old were randomly assigned into four groups in the ratio 2:2:2:1. Children in the first three groups were administered with one dose of live attenuated varicella vaccines manufactured at commercialized scale, and children in the last group were administered with one dose of live attenuated varicella vaccines manufactured at trial-scale .

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 1-3 years old;
* legal identity;
* Guardian(s) of the volunteer should be capable of understanding the written - consent form, and such form should be signed before the children being included into this study.

Exclusion Criteria:

* Prior vaccination with varicella vaccine or with history of varicella infection;
* Axillaty temperature > 37.0 °C before vaccination;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Epilepsy (except febrile seizures), history of seizures or convulsions, a family history of mental illness, autoimmune disease, or immunodeficiency;
* Severe malnutrition, congenital malformation, developmental disorders, or serious chronic diseases;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Receipt of any blood product, immunosuppressant, hormone, other investigational medicine(s) within 30 days prior to study entry;
* Receipt of any live attenuated vaccine within 1 month prior to study entry, or receipt of any subunit vaccine or inactivated vaccine within 7 days prior to study entry;
* Any significant abnormity of heart, lung, liver, spleen, lymph nodes, or pharynx;
* Based on the judgment of investigator(s), there was any condition indicating that the subject should be excluded.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1197 (Actual)
Dates: Start 2014-04-07 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-09-14 (Actual)

PRIMARY OUTCOMES:
The post-immune geometric mean titer (GMT) of susceptible subjects in each group. | 30 days
  Subjects whose pre-immune antibody titer < 1:4 are considered susceptible. The GMT were measured using the method of Fluorescent Antibody to Membrane Antigen (FAMA).
The overall seroconversion rates (SCRs) of each group. | 30 days
  Subjects whose pre-immune antibody titer< 1:4 and post-immune antibody titer≥ 1:4, or those whose pre-immune antibody titer≥1:4 and the increase of post-immune antibody titer≥4 folds are considered seroconverted.

SECONDARY OUTCOMES:
The seroconversion rates (SCRs) of susceptible subjects in each group | 30 days
  Subjects whose pre-immune antibody titer < 1:4 are considered susceptible.
The geometric mean increase (GMI) of susceptible subjects in each group | 30 days
  Increase of post-immune GMT compared with pre-immune GMT.Subjects whose pre-immune antibody titer < 1:4 are considered susceptible.
The overall post-immune GMT of each group | 30 days
  The GMT of all the subjects in each group.
The overall GMI of each group | 30 days
  The GMI of all the subjects in each group.
The incidences of adverse events (AEs) of each group | 30 days
  AEs occurred within 30 days after injection will be collected.
The incidences of serious adverse events (SAEs) of each group | 30 days
  SAEs occurred within 30 days after injection will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Shengli Xia, Principal Investigator — Henan Provincial Center for Disease Control and Prevention